CLINICAL TRIAL: NCT02671201
Title: Training Concepts in Emergency Ultrasonography for Medical Students
Brief Title: Training Concepts in Emergency Ultrasonography
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Cologne (Other)
Responsible Party: Principal Investigator, Guido Michels, Prof. Dr. Guido Michels, University of Cologne
Other Study IDs: 15-412
Record Dates: First submitted 2016-01-27; First posted 2016-02-02 (Estimated); Last update posted 2018-10-17 (Actual); Status verified 2018-10

CONDITIONS: Medical Education in Emergency Ultrasound
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Group A: Theoretical training will be scheduled for 2 hours with lectures in basics of emergency ultrasound. After the theoretical education the students will obtain a bedside-teaching on intensive care unit for 4 hours.
  Interventions: Other: Education
- Group B: Theoretical training will be scheduled for 3 hours and included lectures in echocardiography, lung ultrasound and abdominal ultrasound. After the theoretical education the students will obtain a bedside-teaching on intensive care unit for 3 hours.
  Interventions: Other: Education
- Group C: Theoretical training will be scheduled for 3 hours and included lectures in echocardiography, lung ultrasound and abdominal ultrasound.
  Interventions: Other: Education

INTERVENTIONS:
Other: Education — Different methods in education of emergency ultrasound
  Other Names: Prospective educational study

SUMMARY:
Emergency ultrasound examinations are increasingly important diagnostic tools in emergency and critical care medicine. This study wants to analyze different types of education for undergraduate students. Any method of medical training will be proved theoretical and in clinical practice.

DETAILED DESCRIPTION:
This prospective educational study wants to analyze different methods of education for undergraduate medical students.

Method A: Theoretical training will be scheduled for 2 hours with lectures in basics of emergency ultrasound. After the theoretical education the students will obtain a bedside-teaching on intensive care unit for 4 hours.

Method B: Theoretical training will be scheduled for 3 hours and included lectures in echocardiography, lung ultrasound and abdominal ultrasound. After the theoretical education the students will obtain a bedside-teaching on intensive care unit for 3 hours.

Method C: Theoretical training will be scheduled for 3 hours and included lectures in echocardiography, lung ultrasound and abdominal ultrasound. After the theoretical education the students will obtain a hands-on-training in healthy volunteers for 3 hours. The acquired knowledge and practical skills will be analyzed by a multiple-choice exam (5 MC-questions, 5 video sequences) and a practical exam (five tasks).

Any method of training will be proved at the end theoretical and in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Medical students

Exclusion Criteria:

* No

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Undergraduate medical students
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-06 (Estimated); Primary Completion 2022-01 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Improvement of the knowledge score with different training in emergency ultrasound | 1 year
  With different kinds of short trainings in ultrasound, students can quickly and accurately determine the main emergency ultrasound diagnosis (free fluid, pulmonary consolidation, pulmonary edema, pneumothorax, left and right ventricular failure, pericardial tamponade). The parameter of knowledge score will be used (ratio of multiple choice exam and practical exam).

CONTACTS AND LOCATIONS:
Overall Officials: Guido Michels, Prof. Dr., Study Chair — Univesity of Cologne, Germany
Locations (1):
- Prof. Dr. Guido Michels, Cologne, Germany

IPD SHARING:
Plan to Share IPD: No
No plan to share data.